CLINICAL TRIAL: NCT00446108
Title: Proposal for Retrospective Review of Imaging Pre- and Post - Pulmonary Valve Replacement
Brief Title: Retrospective Pulmonary Valve Replacement Imaging
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Brian Kogon, Associate Professor, Emory University
Other Study IDs: IRB00002765
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Congenital Heart Disease
Keywords: Pulmonary Stenosis; Right Ventricular Dilation; Right Heart Failure; Imaging; Tetralogy of Fallot
MeSH Terms: conditions — Heart Defects, Congenital; Pulmonary Valve Stenosis; Heart Failure; Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective chart review examining children and adults with history of Tetralogy of Fallot or pulmonary stenosis who have undergone subsequent pulmonary valve replacement. The primary interest of the study is to analyze the routine pre- and post-operative imaging studies.

DETAILED DESCRIPTION:
Congenital heart defects having a component of pulmonary stenosis (narrowing) are often palliated in childhood by disrupting the pulmonary valve. This arrangement can provide an excellent quality of life as these children grow and enter young adulthood. Unfortunately, the pulmonary insufficiency that is created by disrupting the pulmonary valve results in volume overload of the right heart. This may eventually lead to right ventricular dilation and irreversible right heart failure. In addition, volume load of the right heart may affect the inter-ventricular septum and left heart function as well. Placement of a competent pulmonary valve at a subsequent operation, hopefully at a time without the replacement valve size constraints present at the initial operation, is a means to eliminate the volume overload and prevent these further sequelae.

Unfortunately, the optimal timing for subsequent pulmonary valve replacement is controversial. One of the currently used indications for valve replacement includes a right ventricular to left ventricular volume ratio greater than two. However, determining the boundaries of the right ventricle by echocardiography and magnetic resonance imaging is difficult in the absence of a pulmonary valve. The boundaries are determined by an arbitrary estimation of where the pulmonary valve should be. Other potential indicators for pulmonary valve replacement may be right ventricular area and right ventricular strain, determined by echocardiography. These measurements are not affected by the absence of the pulmonary valve. They may provide better markers for impending right ventricular failure and a simpler means to follow serial improvement following valve replacement.

While the emphasis after pulmonary valve disruption typically lies on the right ventricle, there is evidence that the left ventricle may become impaired as well. Volume load on the right ventricle causes bowing of the inter-ventricular septum and affects left ventricular function. Echocardiographic imaging of the left ventricle may also be important to follow serial improvement of the left heart following pulmonary valve replacement.

All charts reviewed will be of patients who had their surgery at Children's Healthcare of Atlanta or Emory University Hospital between January 1, 1994 and December 31, 2006. We will review approximately 125 patients' charts for patients between the ages of 1 and 65 years of age who have required pulmonary valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* history of Tetralogy of Fallot or Pulmonary Stenosis
* Pulmonary Valve Replacement
* Surgery at Children's Healthcare of Atlanta or Emory University Hospital between 1.1.94 and 12.31.06
* between 1 and 65 years of age

Exclusion Criteria:

* Those who do not meet inclusion criteria

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a retrospective chart review examining children and adults with history of Tetralogy of Fallot or pulmonary stenosis who have undergone subsequent pulmonary valve replacement. The primary interest of the study is to analyze the routine pre- and post-operative imaging studies. All charts reviewed will be of patients who had their surgery at Children's Healthcare of Atlanta or Emory University Hospital between January 1, 1994 and May 1, 2008. We will review approximately 200 patients' charts for patients between the ages of 1 and 65 years of age who have required pulmonary valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2007-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The first primary aim of the study would be to identify the risk factors for early development of right heart dilation and failure following Tetralogy of fallot repair. | January 1, 1994 and December 31, 2009
  This is a retrospective chart review. The first primary aim of the study would be to identify the risk factors for early development of right heart dilation and failure following Tetralogy of fallot repair.
  The goals would be the following:
  * Determine the risk factors for early pulmonary valve replacement
  * Determine whether there is a positive correlation among the different echocardiographic and MRI parameters
  * Determine whether the parameters improve following pulmonary valve replacement
  * Determine the effects of pregnancy on the right heart
  * Determine the performance of a mechanical valve in the pulmonary position
  * Determine whether the late referral for pulmonary valve replacement worsens patient outcomes
  * Determine whether there is a time of referral beyond which surgery fails to improve patient outcome

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Kogon, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia